CLINICAL TRIAL: NCT03067532
Title: Assessment of Educational Effect of Home-made Robotic Surgery Simulator for Novice Robotic Surgeons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1-2016-0070
Record Dates: First submitted 2017-02-26; First posted 2017-03-01 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Medical School Student; Healthy Population

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental)
  Interventions: Procedure: existed simulation system user
- B (Active Comparator)
  Interventions: Procedure: home made simulator user

INTERVENTIONS:
Procedure: existed simulation system user — Investigator will divide the subject by the two groups. Each group will take about 15 minutes for exercising drive robotic surgery instrument by each simulation system. After 15 minutes, both group will take an short exam to check the ability to manage the robotic surgery instrument.
  Arms: A
Procedure: home made simulator user — Investigator will divide the subject by the two groups. Each group will take about 15 minutes for exercising drive robotic surgery instrument by each simulation system. After 15 minutes, both group will take an short exam to check the ability to manage the robotic surgery instrument.
  Arms: B

SUMMARY:
To overcome the obstacles of endoscopic surgery, the da vinci surgical robot system was applied to the various surgery area . And the complete understanding and practice of the robotic system is very important condition for successful robotic surgery.

Investigator developed a home made robotic surgery simulator for novice robotic surgeons. And investigator want to study about the ability of home made robotic surgery simulator versus existing robotic simulation system.

ELIGIBILITY:
Inclusion Criteria:

1. medical student of Yonsei University College of Medicine
2. first time of robotic surgery system
3. voluntary participation of this study

Exclusion Criteria:

1. minors & foreigner
2. involuntary participation of this study
3. refuse to sign a consent form

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
comparing the understanding and competence level of robotic surgery system | examination day of study participation
  questionnaire : please score the difference after finish this study
  * understanding about the robotic surgery
  * upskilling of the robotic system drive
  * system's advantages
    1. portable
    2. anytime possible
    3. practicality as a real robotic surgery
    4. understandable of using clutch
    5. camera management
  between A and B group system before managing the simulation system and after finishing the simulation system

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No